CLINICAL TRIAL: NCT07290946
Title: Repeated Mesenchymal Stem Cell Therapy for Radiation-Induced Hyposalivation and Xerostomia in Head and Neck Cancer Survivors
Acronym: MESRIX-more
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Christian von Buchwald (Other)
Responsible Party: Sponsor-Investigator, Christian von Buchwald, MD, DMSc, professor, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2025-522559-25-00; 2025-522559-25-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-18; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Xerostomia Due to Hyposecretion of Salivary Gland; Xerostomia Due to Radiotherapy; Sjögren´s Syndrome
Keywords: Mesenchymal Stem Cell; Sjögren; Radiation; xerostomia; Head and Neck cancer
MeSH Terms: conditions — Sjogren's Syndrome; Xerostomia; Head and Neck Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: One research assistant preparing the treatments are unmasked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mesenchymal Stem Cells (Experimental): Treatment with intraglandular injections in both submandibular glands with allogeneic adipose derived mesenchymal stem cells
  Interventions: Drug: ALLOGENEIC AND EXPANDED ADIPOSE TISSUE-DERIVED MESENCHYMAL STEM CELLS
- Placebo (Placebo Comparator): Treatment with intraglandular injections in both submandibular glands sterile isotonic saline water
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALLOGENEIC AND EXPANDED ADIPOSE TISSUE-DERIVED MESENCHYMAL STEM CELLS — Suspended in 10% DMSO. Manufactured by OUH CELL BENCH in Odense, Denmark.
  Arms: Mesenchymal Stem Cells
Drug: Placebo — Sterile isotonic saline water
  Arms: Placebo

SUMMARY:
Dry mouth leads to debilitating symptoms 24/7. The two primary causes for dry mouth are Sjögrens disease and after radiotherapy of a head and neck cancer. Former clinical trials have investigated mesenchymal stem cell treatment for dry mouth with promising results. However, few of the participants evolved normal salivary flow rate. Therefore, in this randomized clinical trial, two treatments of mesenchymal stem cells are administered, 4 months apart. This has not been done before.

The hypothesis is that two treatments of mesenchymal stem cells results in a higher salivary flow rate and ameliorate symptoms from dry mouth.

ELIGIBILITY:
Inclusion Criteria:

1. Former radiotherapy for squamous cell carcinoma, or adenocarcinoma, of the nasal sinus, larynx, pharynx, and oral cavity
2. WHO Performance status 0-1
3. Presence of xerostomia daily
4. UWS of 0.05 mL/min to 0.5 ml/min
5. Age above 18
6. Informed consent
7. 0.5 year follow-up of the cancers in 1. with no recurrence

Exclusion Criteria:

1. Any malignant cancer diagnosis excluding head and neck cancers
2. Xerogenic medications at inclusion
3. Penicillin or streptomycin allergy assessed by health personnel
4. Any other previous or active disease of the salivary glands (e.g. Sjögren's Disease, sialolothiasis)
5. Previous submandibular surgery or biopsy
6. Pregnancy or planned pregnancy until 4 months after second treatment
7. Breastfeeding
8. Smoking within the last 6 months
9. Alcohol abuse within the last 6 months (consumption must not be above 10 units/week (Danish National board health alcohol guidelines)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Unstimulated whole salivary flow rate | T=0 months, T=4 months and T=8 months (primary endpoint assessed after 8 months)
  Unstimulated whole salivary flow rate measured in mL/min

SECONDARY OUTCOMES:
Stimulated whole salivary flow rate | T=0 months, T=4 months, T=8 months (Key secondary endpoint assessed after 8 months).
  Stimulated whole salivary flow rate measured in mL/min
Patient-Reported Outcome of xerostomia: The Groningen Radiotherapy-Induced Xerostomia questionnaire (GRIX). | T=0 months, T=4 months, T=8 months (Key secondary endpoint assessed after 8 months).
  For evaluation of the participants´ perception of xerostomia, the participants will answer validated questionnaires in Danish.
Patient-Reported Outcome of xerostomia: The European organization for research and treatment of cancer quality of life questionnaire, head and neck-35 (EORTC QLQ-H&N35). | T=0 months, T=4 months, T=8 months (Key secondary endpoint assessed after 8 months).
  For evaluation of the participants´ perception of xerostomia, the participants will answer validated questionnaires in Danish. Patients will fill out the EORTC-QLQ- H&N35 (evaluates overall implications of the xerostomia) for the following domains:
  * HNDR: dry mouth
  * HNSS: sticky saliva
  * HNSW: swallowing
Immune response | T=0 months, T=4 months, T=8 months (Key secondary endpoint assessed after 8 months).
  Measured by positivity of de novo drug specific antibodies (binary outcome)
Patient Reported Outcome: Goal Attainment Scale (GAS) | T=0 months, T=4 months, T=8 months (Key secondary endpoint assessed after 8 months).
  Goal attainment Scale (GAS) was developed in 1968 for assessing outcomes in mental health and has since been updated[36]. Now it is used in a wide variety of settings. It is a qualitative patient reported outcome measure. GAS can be beneficial in drug trials where patients have heterogenic symptoms of the disease[37]. The patient, supported by the health professional, picks 3 personal goals to be measured throughout the study period. The goals must be related to the disease and treatment. In this study 3 goals could be: 1. Ability to sleep better at night, ability to eat more solid foods, and less mouth pain. The goals are evaluated at baseline and at each follow up, following the scoring system seen in figure 1. Statistics are calculated from T-scores.

OTHER OUTCOMES:
Incidence of treatment-related adverse events and serious adverse events | Continually assessed from inclusion (T=0 months) to last visit (T=24 months).
  Evaluated by serious adverse events (SAEs), Suspected Unexpected Serious Adverse Reactions (SUSARs), treatment-related adverse events, and deaths.
Outcome 1 to 6 assessed at long term follow-up | T=0 months, T=4 months, T=8 months, T=12 months, and T=24 months
5-point transition scale for determining the minimal important difference (evaluated at 8 months) | T=4 months, T=8 months.
  The 5-point transition scale is critical in the exploratory secondary objective of developing Minimal Important Differences (MIDs) for all the outcome measures applied in the trial because it provides a subjective, patient-centered anchor to assess meaningful change. The scale, which typically ranges from "much worse" to "much better," captures participants' perceptions of change in their condition over time. By linking participants' responses on this scale to corresponding changes in clinical outcome measures, the transition scale helps identify the smallest change in those measures that is considered important or beneficial by the participants themselves. This subjective assessment of change is essential for establishing MIDs, as it ensures that the derived thresholds reflect clinically relevant improvements or deteriorations from the patients' perspectives.

CONTACTS AND LOCATIONS:
Overall Officials: Christian von Buchwald, MD, Professor, Study Chair — Copenhagen University Hospital - Rigshospital

IPD SHARING:
Plan to Share IPD: No
Due to national legislations, few data is anonymized. Therefore, we do not plan to share IPD, unfortunately. However, if it will be possible, this page will be updated.